CLINICAL TRIAL: NCT02123810
Title: Weaker Chest Compression After Nightshift : The We CAN Study.
Brief Title: Quality of Chest Compressions After a Night Shift
Acronym: WeCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bistro Study Group (Other)
Responsible Party: Principal Investigator, Yonathan Freund, Doctor, Bistro Study Group
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BG-CAN
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Arrest
Keywords: fatigue; motor skills; cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Fatigue | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): The investigators measure quality of chest compressions before nightshift. Control group
  Interventions: Other: CPR
- OFF (Other): The investigators measure quality of chest compressions before nightshift. After night shift group
  Interventions: Other: CPR

INTERVENTIONS:
Other: CPR — Simulated cardiac arrest on a manikin Chest Compression CPR for 6 minutes

SUMMARY:
The investigators sought to evaluate the influence of fatigue after a night shift on the quality of Chest Compressions (CC) in CardioPulmonary Resuscitation (CPR), among physicians.

DETAILED DESCRIPTION:
This is a non inferiority cluster randomized trial on three Emergency Departments (ED) and five Intensive Care Unit (ICU) from three urban academic hospital in Paris, France. The investigators evaluated the quality of CC with a low-fidelity manikin and its electronic feedback device. The investigators tested subjects on a 6-minutes CC-only CPR scenario, including 2 minutes of pause. Physicians were tested either on a control day then after a night shift, or after a night shift then on a control day.

ELIGIBILITY:
Inclusion Criteria:

* Resident / Physicians in emergency departement (ED) or taking night in ED
* Resident / Physicians in Intensive Care Unit (ICU) or taking night in ED
* Nightshift > 18 hours

Exclusion Criteria:

* Stop chest compressions before 2 minutes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the proportion of CC with a depth higher than 50mm | 2 minutes of chest compressions
  The investigators evaluated the quality of CC with a low-fidelity manikin and its electronic feedback device.

SECONDARY OUTCOMES:
Number of chest compressions | 2 minutes
  The investigators evaluated the quality of CC with a low-fidelity manikin and its electronic feedback device.

OTHER OUTCOMES:
Factors associated with better chest compressions (CC) | 2 minutes
  The investigators assessed factors associated with better chest compressions as : age, sex and fatigue of physician and intensity of the nightshift.

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, Principal Investigator — Emergency Department, Hôpital Pitié-Salpêtrière, 47-83 Boulevard de l'Hôpital, 75013 Paris, France.
Locations (1):
- Hôpital Pitié-Salpêtrière; Hopital Saint Antoine; Hopital Tenon, Paris, France